CLINICAL TRIAL: NCT06188754
Title: Time-restricted Eating vs. Mediterranean Diet as Adjunctive Interventions for Bipolar Disorder
Brief Title: Healthy Lifestyles for Bipolar Disorder
Acronym: HL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: University College, London (Other); Swinburne University of Technology (Other); Deakin University (Other); University of British Columbia (Other); Salk Institute for Biological Studies (Other); Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Healthy Lifestyles 01
Record Dates: First submitted 2023-12-18; First posted 2024-01-03 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Time Restricted Eating; Diet, Mediterranean
Keywords: bipolar disorder; sleep; circadian rhythm
MeSH Terms: conditions — Intermittent Fasting; Bipolar Disorder | interventions — Diet, Mediterranean

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to take part in either time-restricted eating or the Mediterranean diet.
Who Masked: Outcomes Assessor
Masking Description: Outcomes will be assessed by an interviewer who is unaware of treatment condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time Restricted Eating (TRE) for 8 weeks (Experimental): Participants will receive an intro to TRE and then throughout 8 weeks they will receive brief online psychoeducation several times per week with optional weekly coaching sessions. TRE involves restricting the window of eating to 10 hours/ day, most typically by avoiding eating in the first 1-2 hours after awakening and in the 2-4 before sleep. Those with an eating window > 14 hours will be asked to restrict their eating to 12 hours in the first week, then 10 hours in week 2. To select the period, investigators will ask Ss to review baseline logs to consider sleep, eating, family meals and social commitment schedules, and any special energy demands, such as exercise. During the eating window, no restrictions are placed on the type or quantity of food consumed. The investigators will instruct participants to follow their habitual diet within their 10-hour eating window and to aim to consume the same number of calories per day as they did at baseline.
  Interventions: Behavioral: Time restricted eating
- Mediterranean diet for 8 weeks (Active Comparator): Participants will receive a several page introduction to the mediterranean diet, and then will receive support throughout the 8 week intervention to follow this food plan, including brief online psychoeducation that will be sent several times per week, and optional weekly coaching sessions.
  The mediterranean diet is a plan for healthy eating based on how people eat in the mediterranean region. Individuals will be encouraged to consume vegetables (6 servings/day), fruits (2-4 servings/day), whole grains (daily), legumes (3-4 times per week), nuts (.5 oz per day), and oily fish (2 servings/week). Participants will be encouraged to choose lean meats and other sources of protein over red meat and processed meats. Sweets, refined cereals, alcohol, and wine or alcohol will be labelled as extras, and participants will be encouraged to limit consumption of extras.
  Interventions: Behavioral: Mediterranean diet

INTERVENTIONS:
Behavioral: Time restricted eating — Limiting food intake to 10 hours per day
  Other Names: intermittent fasting
  Arms: Time Restricted Eating (TRE) for 8 weeks
Behavioral: Mediterranean diet — Dietary advice designed to improve consumption of vegetables, fruits, whole grains, and the use of olive oil.
  Arms: Mediterranean diet for 8 weeks

SUMMARY:
The goal of this clinical trial is to compare the effects of two different healthy lifestyles on outcomes for those with bipolar disorder. The goals are to understand the acceptability of time-restricted eating and the mediterranean diet for those who are already receiving medication treatment for bipolar disorder, and to consider how these two food plans predict changes in manic symptoms, depressive symptoms, and Quality of Life. Participants will complete daily measures of eating, sleep and mood for two weeks, and then will be assigned to follow one of the two food plans for eight weeks. The investigators will measure symptoms and Quality of Life at baseline and during and after the food plan.

DETAILED DESCRIPTION:
The investigators will conduct a randomized controlled trial (RCT) to examine the effects of time-restricted eating as compared to the mediterranean diet. In time-restricted eating (TRE), participants will be asked to limit their food intake to a period of 10 hours per day. In the mediterranean diet, participants will be asked to follow a food plan that emphasizes vegetables, fruit, whole grains, and olive oil as central dietary components. The investigators aim to test both food plans as additions to standard medication approaches in bipolar disorder. Participants who are receiving medical treatment for bipolar disorder and who report at least some sleep or circadian problems will complete baseline measures and then will be randomly assigned to TRE or the mediterranean diet for 8 weeks, and then will complete measures of symptoms, Quality of Life, and possible treatment mechanisms at the end of treatment and at 3, 6 and 12 months after the intervention. If successful, this work will provide a novel, easily implemented and highly acceptable intervention for BD.

ELIGIBILITY:
Inclusion Criteria:

* meets diagnostic criteria for bipolar I disorder or bipolar II disorder (but not cyclothymia, BD Not otherwise specified or BD due to another medical condition)
* current sleep (insomnia, hypersomnolence) or circadian sleep-wake (delayed phase, advanced phase, irregular sleep-wake, non-24-hour sleep-wake-type) concerns indicated by endorsement of at least some sleep or circadian-related impairment across the screening self-reports or interview

  * Living in an English-speaking country (and one that we have expertise in research procedures and diet)
  * Has been speaking English for at least 10 years, speaks English in the home, or certifies that they are able to understand English well for the study and demonstrates this during the screening interview.
  * Receiving medical care for BD (referrals will be provided for those who would like to begin care)
  * Mood-stabilizing medication regimens stable for at least one month
  * < 5 kg weight change in the past 3 months
  * Currently eating ≥ 12 hours per day at least twice per week
  * Able to operate the camera function and respond to web-based surveys by phone (loaner phones will be provided as needed)
  * Not engaged in current shift work or have other responsibilities such as providing care that would chronically disrupt their sleep (i.e., > 3 h between 22:00 and 05:00 h for at least 1 day/week)
  * Able to complete 7 days of dietary logs adequately (e.g., at least 2 entries per day, covering at least a 5-hour eating window) during the baseline period
  * Able to complete screening and baseline questionnaires adequately (e.g., not failing more than 1 attention check item with instructed responding; responding to standard multiple-choice items in a mean of < 2 seconds per item). Where individuals respond to more than 14 items in a row with the same response, we will manually review for possible invalidity.

Exclusion criteria include the following:

* Current episode of depression, hypomania or mania, or psychosis (assessed by the aDiagnostic Interview for Anxiety, Mood, and Obsessive-compulsive and Related Neuropsychiatric Disorders; DIAMOND), Participants with acute mood disorder episodes will be encouraged to seek treatment and to consider the study when symptoms have remitted.
* Eating disorder diagnosis (by self-report of treatment or diagnosis at any point during their life, Short Eating Disorder Examination Questionnaire (EDE-QS) scores above clinical concern thresholds for eating disorders, or DIAMOND interview of symptoms during adulthood)
* Past 3-month alcohol use disorder or substance use disorder (assessed by DIAMOND)
* Active suicidal ideation coupled with plan, intent or attempt history as assessed by Columbia Suicide Severity Rating Scale
* Conditions that would interfere with ability to take part in the intervention , including pregnancy, breastfeeding, uncorrected hypo or hyperthyroidism, gastrointestinal conditions impairing nutrient absorption,
* Medical conditions such as HIV, AIDS, lupus, or multiple sclerosis that could confound the assessment of mania or other measures
* Medications contraindicated for fasting: clozapine, glucose-lowering medications, diabetes-related injections, medications requiring food early morning or late evening, corticosteroids; medications such as semaglutide will not be an exclusion criteria
* Cognitive deficits as noted during the initial interview or as indicated by low performance on the Short Orientation Memory Concentration Test (< 20 on the weighted score).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2028-12-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Acceptability | immediately post-treatment (10 weeks after enrollment)
  Participant self-ratings of the acceptability of the intervention: The primary index of acceptability will be the percentage of individuals who endorse that they agree or strongly agree that they would recommend the food plan to a friend. This single item has been used in previous trials of bipolar disorder. Higher agreement will be considered a positive outcome.
Adherence to time-restricted eating | Average number of daily food logs showing adherence across the 8-week intervention
  Adherence will be scored based on the time of their first and final calorie consumption each day during the 8 week intervention. The investigators will select entries from the time interval that contains 95% of intake events. Following standards in other US and European studies of TRE, the investigators will focus on days in which participants adequately logged (e.g., entered at least two intake events, covering at least a 5 hour window), and will calculate the percentage of days in which individuals met the eating window goal. High adherence will be defined as meeting this standard on at least 78% of days logged. As supplemental data, the investigators will report the percentage of days logged, and the percentage of days in which individuals logged adequately and followed the planned window.
Adherence to Mediterranean Diet | Average number of food logs showing adherence at or above the median for 2 days at the mid-point of treatment (week 6) and at the end of treatment (week 10)
  Adherence will be scored based on a Food Frequency Questionnaire that we developed for this study. We will score this using the Adherence to the Mediterranean Diet scoring system (AMed), which provides up to 9 points based on above-median consumption of beneficial foods (e.g., fruits and vegetables) and below median consumption of "extras" such as alcohol. Higher scores reflect better adherence to the mediterranean diet.
Mania | Lower YMRS at the end of intervention (10 weeks) as compared to baseline
  Decline in Young Mania Rating Scale (YMRS) total scores, completed by a blind rater
Depression | Lower MADRS at the end of intervention (10 weeks) as compared to baseline
  Decline in Montgomery Asberg Depression Scale (MADRS) total scores, completed by a blind rater
Self-rated Quality of Life (QOL) | Scores at 1.5-months post-intervention (16 weeks after study entry) as compared to baseline
  Higher scores on the self-rated Brief Quality of Life in Bipolar Disorder (QoL.BD) at 1.5-months post intervention as compared to baseline
Mania at follow-up | YMRS scores will be lower at 3, 6, 12 month post-intervention follow-ups as compared to baseline
  Sustained lower YMRS scores across follow-up
Depression at follow-up | MADRS scores will be lower at 3, 6, 12 month post-intervention follow-ups as compared to baseline
  Sustained lower MADRS scores across follow-up
QOL at follow-up | Brief QOL.BD scores will be higher at 6- and 12-month post-intervention follow-ups as compared to baseline
  Sustained higher Brief QOL.BD scores

SECONDARY OUTCOMES:
Self-rated mania | at post-intervention (10 weeks) and at 1.5, 3, 6, and 12 month follow-ups post-intervention, as compared to baseline
  Lower Patient Health Questionnaire (PHQ) Mania scores at post-intervention (10 weeks) and at 1.5, 3, 6, and 12 month follow-ups post-intervention
Self-rated depression | at post-intervention (10 weeks) and at 1.5, 3, 6, and 12 month follow-ups post-intervention, as compared to baseline
  Lower Patient Health Questionnaire (PHQ) Depression scores at post-intervention (10 weeks) and at 1.5, 3, 6, and 12 month follow-ups post-intervention
Sleep hygiene behaviors | post-intervention (10 weeks) as compared to baseline
  Lower scores on the Sleep Household Environment and In-Bed Behaviors at end-of-treatment (10 weeks) as compared to baseline
Weekly change in mania severity | Weekly scores from the end of the intervention through one-year post-intervention follow-up
  Lower Longitudinal Interval Follow-up Evaluation (LIFE) weekly Mania scores post-treatment as compared to those at baseline. The investigators will administer the LIFE interview at 3, 6, and 12-months after the intervention, and interviewers will record a mania severity rating for each week, to cover the time from the end of intervention until one year after the intervention ends.
Sleep disturbance and sleep impairment | post-treatment (10 weeks) as compared to baseline
  Lower scores on the Patient Outcomes Reporting Information System (PROMIS) sleep disturbance and sleep impairment scores at post-treatment (10 weeks) as compared to baseline
Sleep mid-point variability (Munich Chronotype Questionnaire; MCTQ) | post-treatment (10 weeks) as compared to baseline
  MCTQ scores will show a smaller proportion of individuals with either early or delayed chronotype (as reflected in standard scoring for the MCTQ) at post-treatment as compared to baseline
Regularity of daily routines (Brief Social Rhythm Questionnaire) | post-treatment (10 weeks) as compared to baseline
  Lower Brief Social Rhythm Questionnaire scores (less irregularity) at post-treatment as compared to baseline
Daily emotional lability as assessed using ecological momentary assessment | mid-point of treatment (6 weeks post study entry) as compared to baseline
  Lower mean square of successive difference of negative affect scores within derived from the ecological momentary assessments at the mid-point of treatment (6 weeks) as compared to baseline. Participants will be asked to complete negative affect ratings several times per day for 8 days, at the baseline and mid-point of treatment. The investigators will calculate scores to examine the degree of negative affect variability for each day, and then take the average across 8 days at baseline and at treatment mid-point.

CONTACTS AND LOCATIONS:
Overall Officials: Sheri L Johnson, PhD, Principal Investigator — University of California, Berkeley
Locations (1):
- University of California, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Measures, data, and analysis scripts will be shared through Open Science Foundation.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: De-identified data will be shared within one year after data collection ends.
Access Criteria: Data will be available publically through Open Science Foundation upon request. We will also comply with Wellcome Trust guidance for data sharing.

REFERENCES:
- [Derived] Johnson SL, Murray G, Kriegsfeld LJ, Manoogian ENC, Mason L, Allen JD, Berk M, Panda S, Rajgopal NA, Gibson JC, Joyner KJ, Villanueva R, Michalak EE. A randomized controlled trial to compare the effects of time-restricted eating versus Mediterranean diet on symptoms and quality of life in bipolar disorder. BMC Psychiatry. 2024 May 18;24(1):374. doi: 10.1186/s12888-024-05790-4. PMID 38762486
- Available data/document: Study Protocol — https://pubmed.ncbi.nlm.nih.gov/38762486/